CLINICAL TRIAL: NCT01888211
Title: Effect of Omega 3 Fatty Acid Supplementation on Endothelial Function, Endogenous Fibrinolysis and Platelet Activation in Patients With a Previous Myocardial Infarction
Brief Title: Effect of Omega 3 Fatty Acids on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: LREC/2003/8/13
Record Dates: First submitted 2013-06-12; First posted 2013-06-27 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2013-06

CONDITIONS: Previous Myocardial Infarction
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega 3 fatty acid supplementation (Experimental): Omacor 2 grams daily
  Interventions: Dietary Supplement: Omega 3 fatty acid supplementation
- Olive Oil (Placebo Comparator): Olive Oil capsule 2 grams daily
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acid supplementation — 2 grams Omacor daily
  Arms: Omega 3 fatty acid supplementation
Dietary Supplement: Olive Oil — 2 grams olive oil daily
  Arms: Olive Oil

SUMMARY:
The mechanisms through which omega-3 fatty acids reduce adverse cardiac events remain uncertain. The aim of the study was to investigate the effect of omega-3 fatty acid supplementation on endothelial vasomotor function, endogenous fibrinolysis, and platelet and monocyte activation in patients with coronary heart disease.

DETAILED DESCRIPTION:
Twenty patients with a previous myocardial infarction were recruited into a randomised, double-blind, placebo-controlled, crossover trial of omega-3 fatty acid supplementation (2g/day for 6-weeks). Peripheral blood was taken for analysis of platelet and monocyte activation, and forearm blood flow was assessed in a subset of 12 patients during intrabrachial infusions of acetylcholine, substance P and sodium nitroprusside. Stimulated plasma tissue plasminogen activator (t-PA) concentrations were measured during substance P infusion.

ELIGIBILITY:
Inclusion Criteria:

• Myocardial infarction at least 3 months previously.

Exclusion Criteria:

* Dietary fish allergy or intolerance
* Women of child bearing potential
* Malignant arrhythmias
* Renal or hepatic failure
* Severe or significant co-morbidity
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Lack of informed consent
* Blood donation within last 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Endogenous fibrinolysis (net release of plasma t-PA,IU mL-1) | Measured at 6 weeks after omega 3 fatty acids or placebo
  Endogenous fibrinolysis was measured by drawing blood during intrabrachial substance P infusion and then plasma t-PA antigen and activity (t-PA Combi Actibind Elisa Kit; Technoclone, Vienna, Austria) concentrations were determined by enzyme-linked immunosorbent assays. Estimated net release of plasma t-PA was the product of the infused forearm plasma flow (based on the mean hematocrit and the infused forearm blood flow) and the concentration difference between the infused and noninfused arms.

SECONDARY OUTCOMES:
Endothelial vasomotor function (forearm blood flow, mL l00 mL-1 min-1) | Measured at 6 weeks after omega 3 fatty acids or placebo
  Forearm blood flow was measured during intrabrachial infusions of acetylcholine, substance P and sodium nitroprusside by venous occlusion plethysmography with mercury-in-silicone elastomer strain gauges.
Circulating platelet-monocyte aggregates (%). | Measured at 6 weeks after omega 3 fatty acids or placebo
  Whole blood was immunolabelled with appropriate monoclonal antibodies for subsequent flow cytometric analysis of platelet-monocyte aggregation. Platelet-monocyte aggregates were defined as the percentage of monocytes positive for CD42a.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, Study Chair — University of Edinburgh; Jehangir N Din, Principal Investigator — University of Edinburgh
Locations (1):
- Centre for Cardiovascular Sciences, University of Edinburgh, Edinburgh, Scotland, United Kingdom